CLINICAL TRIAL: NCT06534398
Title: Clinical and Radiographic Outcomes of Implant-supported Prostheses With Cantilever Extensions. A Retrospective Study With a Follow-up of at Least 10 Years.
Brief Title: Clinical and Radiographic Outcomes of Implant-supported Prostheses With Cantilever Extensions After 10 Years of Function
Acronym: Cantilevers
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Other Study IDs: Cantilever implants
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Dental Implants
Keywords: Dental implants; cantilever extension; biologic complications; technical complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Dental implant prosthesis with cantilever extension — A retrospective study on the radiographic and clinical findings of implant-supported dental prostheses with cantilever extensions in place and function for at least 10 years

SUMMARY:
A retrospective examination was performed on patients who had received treatment with dental implants supporting a prosthesis with a cantilever extension for at least 10 years of function.

DETAILED DESCRIPTION:
The successful use of osseointegrated dental implants in replacing missing teeth has been adequately documented, with multiple studies reporting long-term success exceeding 10 years of function. However, there is still insufficient evidence in cases where availability of adequate bone precludes ideal placement of implants. Examples of cases like these include the posterior maxilla when pneumatization of the maxillary sinus does not allow for placement of implants, or areas of thin bone that would require extensive guided bone regeneration (GBR) techniques and increase patient morbidity. In such cases the use of fixed dental prostheses (FDPC's) with cantilever extension has been suggested in lieu of sinus lift techniques or GBR procedures. However, few studies have actually addressed the long-term success of such FDPC's, both from a surgical and a prosthetic standpoint, especially in posterior areas of the mandible and maxilla where loading forces are expected to be higher.

Two studies addressed this issue in the early 2000's with successful outcomes reported for an observation period of 5 years. Others reported similar outcomes after a mean observation period of 5.6 years. The 5th Consensus Conference of the European Association of Osseointegration (EAO) suggested that such treatment can be recommended to patients, albeit with little available evidence and limited follow-up of cases. Recent studies have delved further into this issue, offering longer follow-up data of more than 10 years of function. They included both 2 unit FDP's anchored on one implant and 3 unit FDP's anchored on two implants with cantilever extensions. They concluded that this treatment modality is a reliable option with long-term stability and few complications, mainly prosthetic.

The aim of this retrospective study is to offer further data on the long-term success and complications when at least two dental implants are used to support a FDPC in the posterior areas of both jaws, after at least 10 years of function.

ELIGIBILITY:
The inclusion criteria were as follows:

* Age 18 years and over
* Systemic health or controlled medical conditions
* Periodontal health, either no periodontal disease, or previously treated periodontal disease and under a supportive periodontal maintenance (SPT) program
* Smokers were included but encouraged to enter a smoking cessation program
* Patients with bruxism or parafunctional habits were included.

The exclusion criteria were as follows:

* Uncontrolled medical conditions
* Active uncontrolled periodontal disease
* Inability to present for the reevaluation appointment
* Immediate implant placement
* Cantilever units that were part of full-arch restorations
* Cantilever units that were connected to a single implant
* Non-existent opposing dentition

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patient sample of this study is part of a retrospective evaluation of patients who received treatment with dental implants in a private periodontal practice environment between 2000 and 2013, with at least 10 years of functional loading of their prosthetic work. Patients who received Fixed Dental Prostheses with Cantilever Extension were included in this study sample
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Mean bone loss | 10 years at least
  Mean bone loss measured from the difference of the bone levels at time of implant placement compared to the time of examination

SECONDARY OUTCOMES:
Mean Probing Depth | 10 years at least
  The average probing depth at the time of examination at each implant site
Biologic complications | 10 years at least
  Recording of biologic complications around implants (health, peri-implant mucositis, peri-implantitis
Technical complications | 10 years at least
  Recording of prosthetic complications encountered at the dental prostheses with cantilever extensions

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Vouros, DDS, PhD, Study Chair — Professor of Periodontology
Locations (1):
- Aristotle University of Thessaloniki, School of Dentistry, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wennstrom J, Zurdo J, Karlsson S, Ekestubbe A, Grondahl K, Lindhe J. Bone level change at implant-supported fixed partial dentures with and without cantilever extension after 5 years in function. J Clin Periodontol. 2004 Dec;31(12):1077-83. doi: 10.1111/j.1600-051X.2004.00603.x. PMID 15560808
- [Result] Schmid E, Morandini M, Roccuzzo A, Ramseier CA, Sculean A, Salvi GE. Clinical and radiographic outcomes of implant-supported fixed dental prostheses with cantilever extension. A retrospective cohort study with a follow-up of at least 10 years. Clin Oral Implants Res. 2020 Dec;31(12):1243-1252. doi: 10.1111/clr.13672. Epub 2020 Oct 17. PMID 32991763
- [Result] Aglietta M, Iorio Siciliano V, Blasi A, Sculean A, Bragger U, Lang NP, Salvi GE. Clinical and radiographic changes at implants supporting single-unit crowns (SCs) and fixed dental prostheses (FDPs) with one cantilever extension. A retrospective study. Clin Oral Implants Res. 2012 May;23(5):550-5. doi: 10.1111/j.1600-0501.2011.02391.x. Epub 2012 Jan 17. PMID 22250868
- [Result] Araujo MG, Lindhe J. Peri-implant health. J Periodontol. 2018 Jun;89 Suppl 1:S249-S256. doi: 10.1002/JPER.16-0424. PMID 29926949
- [Result] Baumer A, Toekan S, Saure D, Korner G. Survival and success of implants in a private periodontal practice: a 10 year retrospective study. BMC Oral Health. 2020 Mar 30;20(1):92. doi: 10.1186/s12903-020-01064-z. PMID 32228667
- [Result] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Result] Chappuis V, Buser R, Bragger U, Bornstein MM, Salvi GE, Buser D. Long-term outcomes of dental implants with a titanium plasma-sprayed surface: a 20-year prospective case series study in partially edentulous patients. Clin Implant Dent Relat Res. 2013 Dec;15(6):780-90. doi: 10.1111/cid.12056. Epub 2013 Mar 18. PMID 23506385
- [Result] Derks J, Schaller D, Hakansson J, Wennstrom JL, Tomasi C, Berglundh T. Effectiveness of Implant Therapy Analyzed in a Swedish Population: Prevalence of Peri-implantitis. J Dent Res. 2016 Jan;95(1):43-9. doi: 10.1177/0022034515608832. PMID 26701919
- [Result] Frisch E, Wild V, Ratka-Kruger P, Vach K, Sennhenn-Kirchner S. Long-term results of implants and implant-supported prostheses under systematic supportive implant therapy: A retrospective 25-year study. Clin Implant Dent Relat Res. 2020 Dec;22(6):689-696. doi: 10.1111/cid.12944. Epub 2020 Sep 23. PMID 32969180
- [Result] Gracis S, Michalakis K, Vigolo P, Vult von Steyern P, Zwahlen M, Sailer I. Internal vs. external connections for abutments/reconstructions: a systematic review. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:202-16. doi: 10.1111/j.1600-0501.2012.02556.x. PMID 23062143
- [Result] Halg GA, Schmid J, Hammerle CH. Bone level changes at implants supporting crowns or fixed partial dentures with or without cantilevers. Clin Oral Implants Res. 2008 Oct;19(10):983-90. doi: 10.1111/j.1600-0501.2008.01556.x. PMID 18828813
- [Result] Hammerle CHF, Cordaro L, Alccayhuaman KAA, Botticelli D, Esposito M, Colomina LE, Gil A, Gulje FL, Ioannidis A, Meijer H, Papageorgiou S, Raghoebar G, Romeo E, Renouard F, Storelli S, Torsello F, Wachtel H. Biomechanical aspects: Summary and consensus statements of group 4. The 5th EAO Consensus Conference 2018. Clin Oral Implants Res. 2018 Oct;29 Suppl 18:326-331. doi: 10.1111/clr.13284. PMID 30306690
- [Result] Karoussis IK, Salvi GE, Heitz-Mayfield LJ, Bragger U, Hammerle CH, Lang NP. Long-term implant prognosis in patients with and without a history of chronic periodontitis: a 10-year prospective cohort study of the ITI Dental Implant System. Clin Oral Implants Res. 2003 Jun;14(3):329-39. doi: 10.1034/j.1600-0501.000.00934.x. PMID 12755783
- [Result] Lekholm U, Grondahl K, Jemt T. Outcome of oral implant treatment in partially edentulous jaws followed 20 years in clinical function. Clin Implant Dent Relat Res. 2006;8(4):178-86. doi: 10.1111/j.1708-8208.2006.00019.x. PMID 17100743
- [Result] Mombelli A, van Oosten MA, Schurch E Jr, Land NP. The microbiota associated with successful or failing osseointegrated titanium implants. Oral Microbiol Immunol. 1987 Dec;2(4):145-51. doi: 10.1111/j.1399-302x.1987.tb00298.x. No abstract available. PMID 3507627
- [Result] Pjetursson BE, Zarauz C, Strasding M, Sailer I, Zwahlen M, Zembic A. A systematic review of the influence of the implant-abutment connection on the clinical outcomes of ceramic and metal implant abutments supporting fixed implant reconstructions. Clin Oral Implants Res. 2018 Oct;29 Suppl 18:160-183. doi: 10.1111/clr.13362. PMID 30306682
- [Result] Renvert S, Persson GR, Pirih FQ, Camargo PM. Peri-implant health, peri-implant mucositis, and peri-implantitis: Case definitions and diagnostic considerations. J Periodontol. 2018 Jun;89 Suppl 1:S304-S312. doi: 10.1002/JPER.17-0588. PMID 29926953
- [Result] Roccuzzo M, Bonino L, Dalmasso P, Aglietta M. Long-term results of a three arms prospective cohort study on implants in periodontally compromised patients: 10-year data around sandblasted and acid-etched (SLA) surface. Clin Oral Implants Res. 2014 Oct;25(10):1105-12. doi: 10.1111/clr.12227. Epub 2013 Jul 19. PMID 23865554
- [Result] Romeo E, Tomasi C, Finini I, Casentini P, Lops D. Implant-supported fixed cantilever prosthesis in partially edentulous jaws: a cohort prospective study. Clin Oral Implants Res. 2009 Nov;20(11):1278-85. doi: 10.1111/j.1600-0501.2009.01766.x. Epub 2009 Aug 26. PMID 19709064
- [Result] Storelli S, Del Fabbro M, Scanferla M, Palandrani G, Romeo E. Implant-supported cantilevered fixed dental rehabilitations in fully edentulous patients: Systematic review of the literature. Part II. Clin Oral Implants Res. 2018 Oct;29 Suppl 18:275-294. doi: 10.1111/clr.13310. PMID 30306687